CLINICAL TRIAL: NCT07311057
Title: Investigation of Effect of Formulated Methylene Blue on Treatment of Squamous Cell Carcinoma Skin Cancer in Inoperable Patients and Not Suitable for Radiotherapy
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Daryoush Hamidi Alamdari, PhD (Other)
Responsible Party: Sponsor-Investigator, Daryoush Hamidi Alamdari, PhD, Professor, Mashhad University of Medical Sciences
Organization: Mashhad University of Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IR.MUMS.IRH.REC.1404.226
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: SCC - Squamous Cell Carcinoma; SCC - Squamous Cell Carcinoma of Skin; Inoperable Disease
Keywords: Squamous cell carcinoma; Methylene blue; Carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Formulated Methylene Blue Treatment Arm (Experimental): Participants in this single-arm, open-label pilot study will receive topical methylene blue-based dressing for the management of advanced or inoperable squamous cell carcinoma (SCC) wounds. Wound area and depth will be evaluated weekly for four weeks using standardized digital photography (30 cm distance) and sterile metallic measurement tools. Images will be analyzed with HealUp software to quantify wound area and healing progression. The study aims to preliminarily assess the efficacy and safety of methylene blue in promoting wound healing among five patients with refractory SCC lesions who are not candidates for surgery or radiotherapy.
  Interventions: Drug: Formulated Topical Methylene Blue (0.5 mg/mL); Drug: Wound Healing Gel

INTERVENTIONS:
Drug: Formulated Topical Methylene Blue (0.5 mg/mL) — Participants will receive a topical formulation of methylene blue at a concentration of 0.5 mg/mL, applied directly to the squamous cell carcinoma (SCC) lesions. The formulation will be administered every two days for a period of one month. The topical preparation is designed with a standard cream base containing carrier oils and lipids to enhance penetration into deeper skin layers and facilitate the delivery of the active compound. Additional excipients include zinc oxide and copper to support wound healing. Clinical photographs of the lesions will be taken at each application to monitor treatment progress.
Drug: Wound Healing Gel — Following completion of the methylene blue treatment, a wound healing gel will be applied to the treated lesions. This gel, which contains platelet-rich fibrin and other supportive compounds, has demonstrated efficacy in removing necrotic tissue and promoting tissue regeneration. The gel will be used until complete wound closure is achieved.

SUMMARY:
The goal of this clinical trial is to evaluate whether formulated methylene blue can safely and effectively treat advanced or inoperable Squamous Cell Carcinoma (SCC), a common type of skin cancer. This condition mainly affects adults and often occurs on the head or neck. Some patients cannot undergo surgery or radiotherapy due to tumor invasion, recurrence, or health limitations.

The main questions this study aims to answer are:

Can formulated methylene blue reduce tumor size and promote healing in patients with advanced SCC? Is this treatment safe and well-tolerated? There is no comparison group in this study. Researchers will assess each patient's response before and after the treatment.

Participants will:

Receive topical methylene blue solution or ointment applied to the affected skin every two days for one month.

Undergo clinical and photographic evaluation before, during, and after treatment.

Use a proven wound-healing gel following methylene blue therapy to assist tissue recovery.

Blood tests and clinical follow-up will be conducted for six months to monitor safety and long-term effects. The study aims to provide new evidence for a non-invasive and low-cost therapeutic option for patients who cannot receive standard treatments.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed diagnosis of squamous cell carcinoma (SCC)
* Provision of written informed consent to participate in the study
* Lack of willingness or eligibility for surgical excision or radiotherapy, or contraindication to intralesional medical treatments such as interferon-alpha or 5-fluorouracil (5-FU)
* Age ≥ 18 years
* Lesion size < 2 cm in diameter
* Presence of multiple lesions

Exclusion Criteria:

* Withdrawal of consent at any stage of the study
* Pregnancy or breastfeeding
* History of severe adverse reactions to medications
* Inability or unwillingness to attend follow-up visits
* History of cardiovascular disease
* History of thromboembolic disorders
* Prior radiotherapy to the affected area
* History of chronic arsenic exposure
* Immunodeficiency
* Presence of severe systemic illness
* Known allergy or hypersensitivity to methylene blue
* History of bleeding disorders or abnormal coagulation
* Severe inflammatory or dermatologic conditions in the treatment area
* Failure to complete the full course of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-20 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Rate of Wound Healing and Tumor Regression in Inoperable squamous Cell Carcinoma Treated with Topical Formulated Methylene Blue | Baseline, every week for 4 weeks during treatment, and at 8 weeks post-treatment follow-up.
  The primary outcome of this study is to evaluate the efficacy of topical formulated methylene blue (0.5 mg/mL) in promoting wound healing and reducing tumor size in patients with inoperable or radiotherapy-resistant squamous cell carcinoma (SCC). The assessment includes measurement of wound area and depth using standardized digital photography and calibrated sterile metal measurers. Images will be analyzed with the HealUp software to determine the rate of epithelialization and reduction in lesion size. The degree of tissue regeneration and clinical response will be documented before treatment and at defined follow-up intervals.

SECONDARY OUTCOMES:
Changes in Inflammatory and Biochemical Markers Before and After Treatment with Topical Formulated Methylene Blue | At baseline (before treatment) and at completion of therapy (approximately 4 to 8 weeks after treatment initiation).
  The secondary outcome is to assess the variation in systemic inflammatory and biochemical parameters, including C-reactive protein (CRP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST), measured before initiation of treatment and after complete wound healing. These biomarkers will be evaluated to determine the systemic safety profile and potential anti-inflammatory effects of topical formulated methylene blue. Blood samples will be analyzed in the central laboratory of Imam Reza Hospital using standard clinical chemistry assays.

CONTACTS AND LOCATIONS:
Locations (1):
- Mashhad University of Medical Sciences, Mashhad, Khorasan Razavi, Iran

IPD SHARING:
Plan to Share IPD: No